CLINICAL TRIAL: NCT04775641
Title: Children and Neonates Anaesthesia in Magnetic Resonance Environment in Italy. An Active Call Survey
Brief Title: Italian Survey on Paediatric and Neonatal MRI
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, SPINAZZOLA GIORGIA, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: MRI001
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Cerebral Disorders Congenital; Premature Birth
MeSH Terms: conditions — Premature Birth | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionnaire — questionnaire

SUMMARY:
Paediatric anaesthesia care in the Magnetic Resonance Imaging is a challenge for clinicians. The recent debate about the role of anaesthetic agent on neural development, encouraged an evaluation of their actual activity in this environment. In this active call survey, the authors sought to delineate the Italian situation regarding national centers, staff involved, monitoring and tools available. The primary aim was to evaluate clinical practice in childhood management in Magnetic Resonance suite.

This study was designed as prospective phone survey on the setting of a complete sample of all national centers performing almost a paediatric discharge in the 2014, obtained from Italian Health Ministery registers.

The three section survey was fill out with the Physician in charge in Magnetic Resonance suite. The Main outcome was a descriptive and exploratory analyses about the organization setting of the Centers (procedures, performers, monitoring and tools).

ELIGIBILITY:
Inclusion Criteria:

* Uncooperative children < 14 years old
* premature babies

Exclusion Criteria:

. collaborating children

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All center perforing a paediatric discharge in Italy in the 2014
Sampling Method: Non-Probability Sample
Enrollment: 876 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Descriptive practice for children and neonates management in MRI | 3 monthes

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Gemelli, Rome, Italy

REFERENCES:
- [Derived] Sbaraglia F, Spinazzola G, Adduci A, Continolo N, De Riso M, Ferrone G, Festa R, Garra R, Tosi F, Rossi M. Children and neonates anesthesia in magnetic resonance environment in Italy: an active call survey. BMC Anesthesiol. 2022 Sep 2;22(1):279. doi: 10.1186/s12871-022-01821-3. PMID 36056321